CLINICAL TRIAL: NCT06505980
Title: Stop, Focus, Plan, and Change: A Translational Approach to Predict Parent and Child Responses to a Brief, Telehealth Parent Training
Brief Title: Stop, Focus, Plan, and Change: Predicting Parent and Child Responses to a Brief, Telehealth Parent Training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-3184; 1K23MH134189-01A1 (NIH)
Record Dates: First submitted 2024-06-18; First posted 2024-07-17 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Behavioral Problem; Irritable Mood; Parenting; Stress
Keywords: Behavioral Concerns; Irritability; Parenting stress; Parenting practices
MeSH Terms: conditions — Problem Behavior

STUDY DESIGN:
Masking Description: Coders will be masked to treatment time-point when measuring observed outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Parent Training Program (Other): The behavioral parent training intervention is delivered briefly through telehealth. It will be the only arm. It will be the only intervention received by participants in the context of this study.
  Interventions: Behavioral: Brief Behavioral Parenting Program

INTERVENTIONS:
Behavioral: Brief Behavioral Parenting Program — The brief behavioral parenting program is a 6 session, group-based behavioral parent training program. The components include support-building, parenting strategy education, and actively practicing parenting strategies. It is delivered through telehealth.
  Other Names: Behavioral Parent TRaining

SUMMARY:
This study will look at who does not improve after doing a behavioral parent training program briefly through telehealth. It will also study ways to make the intervention better for those that do not improve.

ELIGIBILITY:
Inclusion Criteria:

* Parent speaks English or Spanish
* Parent has access to Internet
* Parent intends to complete treatment
* Parent reports child has elevated externalizing concerns

Exclusion Criteria:

* Child is a ward of the state
* Child diagnosed with severe medical or nonverbal developmental disability

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 130 (Estimated)
Dates: Start 2024-10-18 (Actual); Primary Completion 2028-11-01 (Estimated); Study Completion 2029-03-30 (Estimated)

PRIMARY OUTCOMES:
Parenting Scale - Short Form | (1) Pre-treatment, (2) Up to 4 weeks after treatment began (Mid-Treatment), and (3) Up to 12 weeks after treatment began (Post-treatment)
  The Parenting Scale Short Form measures parenting practices, including emotional over-reactivity and lax discipline use. Possible scores on the emotional over-reactivity scale range from 4 to 28, with higher scores indicating more emotional reactivity. Possible scores on the lax discipline scale range from 4 to 28, with higher scores indicating more lax discipline use.
Caregiver Strain Questionnaire - Short Form | (1) Pre-treatment, (2) Up to 4 weeks after treatment began (Mid-Treatment), and (3) Up to 12 weeks after treatment began (Post-treatment)
  The Caregiver Strain Questionnaire - Short Form measures parenting stress. Possible scores range from 7 to 35, with higher scores indicating more parenting stress.
Eyberg Child Behavior Inventory | (1) Pre-treatment, (2) Up to 4 weeks after treatment began (Mid-Treatment), and (3) Up to 12 weeks after treatment began (Post-treatment)
  The Eyberg Child Behavior Inventory measures parent-reported child behavioral concerns. Possible scores range from 36 to 252, with higher scores indicating more child behaviors concerns.
Sutter Eyberg Student Behavior Inventory | (1) Pre-treatment and (3) Up to 12 weeks after treatment began (Post-treatment)
  The Sutter Eyberg Student Behavior Inventory measures teacher-reported child behavioral concerns. Possible scores range from 36 to 266, with higher scores indicating more child behaviors concerns.

SECONDARY OUTCOMES:
PROMIS Child Anger / Irritability | (1) Pre-treatment, (2) Up to 4 weeks after treatment began (Mid-Treatment), and (3) Up to 12 weeks after treatment began (Post-treatment)
  The PROMIS Child Anger / Irritability survey measures child irritability. Possible scores range from 8 to 40, with higher scores indicating more child irritability.
Parent-Child Interaction Coding System | (1) Pre-treatment and (3) Up to 12 weeks after treatment began (Post-treatment)
  The Parent-Child Interaction Coding System (PARCHISY) is an observational coding system measuring parenting behavior and affect. Observation are coded using global ratings on a 1 (not observed) to 7 (frequently observed) scale.
Dyadic Parent-Child Interaction Coding System | (1) Pre-treatment and (3) Up to 12 weeks after treatment began (Post-treatment)
  The dyadic parent-child interaction coding system is an observational coding system measuring parenting behaviors. Observations are coding using event-based ratings to tally the number of specific parenting behaviors observed within the parent-child interaction task.
Retrospective Post-Pre Change: Harsh Parenting | (3) Up to 12 weeks after treatment began (Post-treatment)
  The retrospective post-pre change: harsh parenting questionnaire measures parental perceptions of change in harsh parenting (e.g., yelling) over the course of the intervention. One item measures the frequency of harsh parenting before the intervention and another item measures the frequency of harsh parenting after the intervention. Each item ranges from 0 to 100 with higher scores indicating more harsh parenting at the respective time point.
Retrospective Post-Pre Change: Parenting Stress | (3) Up to 12 weeks after treatment began (Post-treatment)
  The retrospective post-pre change: parenting stress questionnaire measures parental perceptions of change in parenting stress over the course of the intervention. One item measures the frequency of parenting stress before the intervention and another item measures the frequency of parenting stress after the intervention. Each item ranges from 0 to 100 with higher scores indicating more parenting stress at the respective time point.
Retrospective Post-Pre Change: Child Externalizing Concerns | (3) Up to 12 weeks after treatment began (Post-treatment)
  The retrospective post-pre change: child behavioral concerns questionnaire measures parental perceptions of change in child behavioral concerns over the course of the intervention. One item measures the frequency of child behavioral concerns before the intervention and another item measures the frequency of child behavioral concerns after the intervention. Each item ranges from 0 to 100 with higher scores indicating more child behavioral concerns at the respective time point.
Retrospective Post-Pre Change: Child Irritability | (3) Up to 12 weeks after treatment began (Post-treatment)
  The retrospective post-pre change: child irritability questionnaire measures parental perceptions of change in child irritability over the course of the intervention. One item measures the frequency of child irritability before the intervention and another item measures the frequency of child irritability after the intervention. Each item ranges from 0 to 100 with higher scores indicating more child irritability at the respective time point.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States